CLINICAL TRIAL: NCT03159494
Title: A Self-monitoring Approach in Evaluating the Effect of 3 Weeks of High-Intense Interval Training in Type 2 Diabetics
Brief Title: High-intensity Training, Self-monitoring and Diabetes 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOU-PHD-007
Record Dates: First submitted 2017-05-02; First posted 2017-05-18 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus; High-Intensity Interval Training; Self Care
MeSH Terms: conditions — Diabetes Mellitus | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A pilot group of 6 patients with type 2 diabetes tested before and after 6 times of High Intensity Training One group of patients with type 2 diabetes tested before and after 8 times of High Intensity Training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 10 patients with type 2 diabetes enrolled to perform 8 times of High-Intensity Training. The subjects were tested before and after the training period.
  Interventions: Other: High-Intensity Training
- Pilot study (Experimental): 6 patients with type 2 diabetes enrolled to perform 6 times of High-Intensity Training. The subjects were tested before and after the training period
  Interventions: Other: High-Intensity Training

INTERVENTIONS:
Other: High-Intensity Training — 8 times of Hit consisting of 3 minutes of Warm-up on an indoor bike followed by 10 intervals of 1 minute at 90% og HRmax interspersed of 1 minute of recovery.
  As for the pilot study 6 times of training were completed

SUMMARY:
10 patients with type 2 diabetes participated in a training-intervention consisting of 8 times of High-Intensity Training (HIT). Before and after the intervention the patients were tested regarding Oral Glucose Tolerance Test, blood pressure, weight and fat% and VO2max. A pilot study was conducted with 6 patients with type 2 diabetes using the same protocol but only 6 times of training.

DETAILED DESCRIPTION:
The aim of the study is to investigate to which extent a short period of HIT can improve cardio-metabolic status measured by simple methods such as OGTT (fasting glucose and 2h-glucose), blood pressure, weight and fat percent in patients with type 2 diabetes

Protocol:

At day -2 a VO2max test was performed in order to get familiarized to the test before the actual test at day 0. The pretest at day 0 was carried out at least two days before the first training session in order to allow patients to recover after the Vo2max test before training. After 8 times of training the posttest was accomplished at day 21 two days after the last training session in order to avoid the acute effect of training. Both pre- and posttest were carried out on Fridays and training days were Mondays, Wednesdays and Fridays.

The pre- and posttest contained the following: Oral glucose tolerance test (OGTT), blood pressure measurement, weight and fat% measurements and VO2maxtest. Pretesting also contained a questionnaire about physical activity and their medical history in addition to the physiological tests.

Oral Glucose Tolerance Test (OGTT): Participants were instructed to continue a normal diet in the days leading up to the test. At the day of testing they should meet fasting (for at least 10 hours) and they were asked not to take any medications that could influence blood glucose levels in the fasting hours (two forgot and they were instructed also to take medications prior to the posttest). At baseline a small blood sample was collected by the use of a finger prick to determine fasting capillary blood glucose level (producent). The fingertip was disinfected before the finger prick and the first drop of blood was removed before applying a drop of blood in the glucose meter. The participants were then instructed to drink 75 mg of glucose dissolved in 300 ml of water. Blood samples were collected after 30, 60, 90 and 120 minutes with the use of finger prick.

Blood pressure: Blood pressure was measured after 10 min of rest in a sitting position. An automatic blood pressure monitor was used (producent) and three measures were made. The lowest of the three values were used in calculations.

Weight and fat%: Weight and fat% were measured on a Tanita digital scale with bioelectrical impedance. The participants were instructed to step on the scale barefooted and to keep the hands with the handgrips slightly elevated from the torso.

VO2max: Bicycle test on a Lode ergometer bike to exhaustion with direct measurement of oxygen consumption by Breath-by-breath on Masterscreen CPX. The participants were instructed about the protocol before applying the equipment used for the test. Then there was a warm-up for 5 min. on 50-75 watt followed by incremental increase in intensity by 25 watt each minute until exhaustion. The test was considered a VO2max if the RER-value exceeded 1,10. Otherwise, is was categorized as a VO2peak test.

Physical activity: Physical activity was assessed by using the Physical Activity Scale (PAS) questionnaire (19). PAS1 was used instead of the PAS2 as not all the participants were working in the daytime. The participants were asked to report time spend on different activities on an average weekday before the intervention. These activities are categorized into nine different categories with a corresponding metabolic equivalent (1 MET ~1 kcal/kg/h) ranging from low to high intensity. A total MET-score was calculated as time spend on each category multiplied by the corresponding MET and then all nine categories were added together. The categories are sleep (0.9 MET), TV-viewing/reading (1.0 MET), sitting/working (1.5 METs), standing up (2.0 METs), light work (3.0 METs), light to moderate activity (4.0 METs) moderate activity (5.0 METs), moderate to high activity (6.0 METs) and high intensity activity (>6 METs). As for the high intensity 7 METs was chosen in this study.

Training: The training consisted of 10 x 60 sec work on an indoor exercise bike at an intensity of ~90% of max HR interspersed by 60 sec of recovery 3 times per week (Mon-Wed-Fri) with a total amount of eight training sessions. This protocol was the same as used by Little et al (2011). The pedal cadence was individually set in the area of 80 -110 rpm. In the recovery the participants pedalled slowly at a lower intensity (~ 50 watt). The HR used for training was calculated based on the max HR found by VO2max test at pretest. Each interval was scored on Borg Scale (rate of perceived exhaustion, RPE) which is a subjective scale where the participants experience of exhaustion is expressed in a number from 6 to 20. 14-15 is determined as where speaking in sentences is interrupted by breath and at 16-17 there is a clear hyperventilation. Perceived enjoyment of low-volume HIT was assessed by asking participants how enjoyable they would find engaging in 1) a single bout of HIT (10 x 1 min) and 2) HIT at least 3 times/wk for the next 4 wk using a 9-point Likert scale ranging from 1 (not enjoyable at all) to 9 (very enjoyable).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 diabetes
* Approved to participate by own general practitioner

Exclusion Criteria:

* Conditions contraindicating training at high intensity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2015-11-13 (Actual); Study Completion 2015-11-13 (Actual)

PRIMARY OUTCOMES:
Fasting glucose concentration | Through study completion, an average of 3 weeks
  A small blood sample was collected by the use of a finger prick to determine fasting capillary blood glucose level (mmol/l) by a glucose meter (Accu Check)
2-hour glucose concentration | Through study completion, an average of 3 weeks
  The participants were instructed to drink 75 mg of glucose dissolved in 300 ml of water. Blood samples were collected after 30, 60, 90 and 120 minutes with the use of finger prick and blood concentrations were measured by a glucose meter (Accu Check)
Weight | Through study completion, an average of 3 weeks
  Weight measured i kilograms on a Tanita digital scale without shoes
Fat percent | Through study completion, an average of 3 weeks
  A Tanita digital scale with bioelectric impedance was used to measured fat percent (%)
Oxygen consumption | Through study completion, an average of 3 weeks
  Bicycle test on a Lode ergometer bike to exhaustion with direct measurement of oxygen consumption by Breath-by-breath on Masterscreen CPX. The participants were instructed about the protocol before applying the equipment used for the test. Then there was a warm-up for 5 min. on 50-75 watt followed by incremental increase in intensity by 25 watt each minute until exhaustion. The outcome was measured in l/min and ml/kg/min
Training intensity | Through study completion, an average of 3 weeks
  The training intensity measured i % of max heart rate and Borg´s rate of perceived exhaustion was made for each interval (10 intervals/training, 8 times of training)
Blood pressure | Through study completion, an average of 3 weeks
  Blood pressure was measured after 10 min of rest in a sitting position. An automatic blood pressure monitor was used and three measures were made. The lowest of the three values were used in calculations.

SECONDARY OUTCOMES:
Physical acitity | At baseline
  The participants level of physical activity (measured in MET´s) was calculated by the use of the Physical Activity Scale (Aadahl M & Joergensen T, 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Ole K Hejlesen, Professor, Principal Investigator — Medical Informatics, Aalborg University, Denmark

IPD SHARING:
Plan to Share IPD: No